CLINICAL TRIAL: NCT02128646
Title: Liposomal Bupivacaine (Exparel) for Postoperative Pain Control for Open and Laparoscopic Abdominal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000101
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: Pain Management; Exparel; Abdominal Hernia Repair; Laparoscopic Surgery
MeSH Terms: conditions — Pain; Agnosia | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Group 1 (Experimental): Treatment Group patients will receive an opioid-sparing, multimodal, postsurgical pain regimen consisting of intraoperative local wound infiltration with 266 mg EXPAREL followed by, when not contraindicated, administration of a 30 mg dose of IV ketorolac at the end of surgery. Patients scheduled in Treatment Group 1 will have an open surgery for abdominal hernia repair.
  Interventions: Drug: EXPAREL; Drug: Ketorolac; Procedure: an open surgery for abdominal hernia repair
- Treatment Group 2 (Experimental): Treatment Group patients will receive an opioid-sparing, multimodal, postsurgical pain regimen consisting of intraoperative local wound infiltration with 266 mg EXPAREL followed by, when not contraindicated, administration of a 30 mg dose of IV ketorolac at the end of surgery. Patients scheduled in Treatment Group 2 will have a laparoscopic abdominal hernia repair.
  Interventions: Drug: EXPAREL; Drug: Ketorolac; Procedure: laparoscopic abdominal hernia repair
- Control Group 1 (Active Comparator): Patients scheduled in Control Group 1 will have an open surgery for abdominal hernia repair. The Control Group patients will receive traditional treatment.
  Interventions: Procedure: an open surgery for abdominal hernia repair
- Control Group 2 (Active Comparator): Patients scheduled in Control Group 2 will have laparoscopic abdominal hernia repair. The Control Group patients will receive traditional treatment.
  Interventions: Procedure: laparoscopic abdominal hernia repair

INTERVENTIONS:
Drug: EXPAREL
  Other Names: Bupivacaine Liposome Injectable Suspension
  Arms: Treatment Group 1; Treatment Group 2
Drug: Ketorolac
  Other Names: Toradol
  Arms: Treatment Group 1; Treatment Group 2
Procedure: laparoscopic abdominal hernia repair
  Arms: Control Group 2; Treatment Group 2
Procedure: an open surgery for abdominal hernia repair
  Arms: Control Group 1; Treatment Group 1

SUMMARY:
The purpose of this study is to learn how well Liposomal Bupivacaine (Exparel™) controls post-operative pain in patients undergoing both open and laparoscopic (minimally invasive) abdominal hernia repair surgery.

DETAILED DESCRIPTION:
When a person has surgery, there are a few different standard care options for pain relief. Anesthetic (numbing) drugs can be used to cause a loss of feeling in or around a wound but the effect of the numbing medication can be undone.Pain relieving drugs such as acetaminophen (Tylenol), non-steroidal anti-inflammatory drugs (NSAIDs), and opioid (narcotic) medications can also be taken by mouth or through a vein in your arm (intravenous IV.) However, both NSAIDs & Opioid drugs can produce negative side effects such as serious difficulty breathing, stopping breathing altogether, low blood pressure, nausea, vomiting, itching, and constipation.

Bupivacaine is one of the commonly used longer-acting numbing medicines (anesthetics). The effect of Bupivacaine or other anesthetics is limited to usually no more than 12 hours when injected around the area of the incision during surgery. Liposomal Bupivacaine (Exparel) could provide good, continuous and longer pain relief than current therapies/treatments commonly used. This can possibly improve patient satisfaction and time to normal activities such as walking.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo an open or laparoscopic abdominal hernia repair.
* Ability to provide informed consent, adhere to study visit schedule, and complete all study assessments.

Exclusion Criteria:

* Patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioids or ketorolac.
* Patients who abuse alcohol or other drug substance.
* Patients who are on chronic opioid therapy (taken an opioid 5 of the last 7 days).
* Patients with severe hepatic impairment.
* Patients currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Moncure, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Laparoscopic Treatment Arm: Laparoscopic abdominal hernia repair with Exparel
- Laparoscopic Control Arm: Laparoscopic abdominal hernia repair without Exparel
- Open Treatment Arm: Open abdominal hernia repair with Exparel
- Open Control Arm: Open abdominal hernia repair without Exparel
Period: Overall Study
Arm/Group | Laparoscopic Treatment Arm | Laparoscopic Control Arm | Open Treatment Arm | Open Control Arm
Started | 7 | 4 | 5 | 3
Completed | 7 | 4 | 5 | 2
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Laparoscopic Treatment Arm; Laparoscopic Control Arm: All patients 18 and older presenting with an abdominal hernia requiring laparoscopic repair were screened for inclusion.
- Open Treatment Arm; Open Control Arm: All patients 18 and older presenting with an abdominal hernia requiring open surgical repair were screened for inclusion.
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Treatment Arm | Laparoscopic Control Arm | Open Treatment Arm | Open Control Arm | Total
Number analyzed (Participants) | 7 | 4 | 5 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 2 | 2 | 11
  >=65 years | 3 | 1 | 3 | 1 | 8
Age, Continuous [Median (Full Range); unit: years] — Population: Different arms have different age ranges and number of participants.
  years | 60.5 [38 to 83] | 62 [47 to 77] | 74.5 [59 to 90] | 55.5 [41 to 70] | 64 [38 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 4
  Male | 5 | 3 | 5 | 2 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 4 | 5 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With Pain Management After Surgery
Description: Satisfaction measured with composite score that includes score from the Likert scale and opioid consumption/satisfaction log. Satisfaction was rated on a scale of 1-5, with 1 being "strongly disagree"/not satisfied with pain control and 5 being "strongly agree"/satisfied with pain control. Patients filled out the log on days 1-4 after surgery and at a 7-14 day follow up visit.
Time Frame: Change from Surgery to Day 14
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Laparoscopic Control Arm; Open Control Arm: Patients were eligible for opioid treatment during surgery and did not receive Exparel.
- Laparoscopic Treatment Arm; Open Treatment Arm: Patients may have received Fentanyl during surgery, but all other opioids were prohibited. They all received 266 mg of Exparel, followed by 30 mg of IV Ketorolac when not contraindicated.
Arm/Group | Laparoscopic Control Arm | Laparoscopic Treatment Arm | Open Control Arm | Open Treatment Arm
Number analyzed (Participants) | 4 | 7 | 2 | 5
score on a scale | 4 [3.5 to 4] | 4 [4 to 5] | 2.5 [2 to 3] | 5 [4 to 5]

2. Secondary Outcome: Total Length of Time in Post-anesthesia Care Unit (PACU)
Description: Length of time subjects stayed in the PACU following surgery
Time Frame: Up to 385 minutes after surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Open Control; Laparoscopic Control: Patients were eligible for opioid treatment during surgery and did not receive Exparel.
- Open Treatment; Laparoscopic Treatment: Patients may have received Fentanyl during surgery, but all other opioids were prohibited. They all received 266 mg of Exparel, followed by 30 mg of IV Ketorolac when not contraindicated.
Arm/Group | Open Control | Open Treatment | Laparoscopic Control | Laparoscopic Treatment
Number analyzed (Participants) | 2 | 5 | 4 | 7
minutes | 93.5 [69 to 118] | 64 [60 to 93] | 118 [76.5 to 151] | 86 [55 to 98]

ADVERSE EVENTS:
Time Frame: Patients were assessed for AE/SAE daily while inpatient and then through patient report during the 7-14 day follow-up visit.
Groups:
- Open Control Arm; Open Treatment Arm; Laparoscopic Control Arm; Laparoscopic Treatment Arm: Patients were assessed for AE/SAE daily while inpatient and then through patient report during the 7-14 day follow-up visit.
Arm/Group | Open Control Arm | Open Treatment Arm | Laparoscopic Control Arm | Laparoscopic Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/4 | 0/7

LIMITATIONS AND CAVEATS:
Trial was ended prematurely due to administrative constraints and only reached half of the projected enrollment numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No